CLINICAL TRIAL: NCT01235832
Title: The Effect of One Avocado Per Day on Established and Emerging Cardiovascular Disease (CVD) Risk Factors
Brief Title: The Effect of Avocado on Cardiovascular Disease (CVD) Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PKE 106
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease; Hyperlipidemia
Keywords: cholesterol; triglycerides; low-density lipoprotein; high-density lipoprotein; reverse cholesterol transport
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lower-Fat Diet (Active Comparator): The Lower-Fat diet will provide ~24% of calories from fat and meet the SFA and cholesterol recommendations of a Step-II diet recommended by the National Heart, Lung, and Blood Association's National Cholesterol Education Program. SFA will provide 7% of calories, and cholesterol will be less than 200mg/day. Vegetables and fruits in the Lower-Fat diet will be selected from foods that are low in antioxidants.
  Interventions: Other: Lower-Fat Diet
- Moderate Fat Diet (Active Comparator): This diet is designed to be the control diet for the avocado diet and will have an identical fatty acid profile. MUFA-enriched food (fats) will be substituted for avocado. The substitution foods will not contain antioxidant or cholesterol-lowering components similar to those in avocado.
  Interventions: Other: Moderate Fat Diet
- Avocado Diet (Experimental): The avocado diet will be designed to ensure that all subjects incorporate 1 avocado (~136g) per day into a moderate fat diet. Both the Lower-Fat diet and avocado diet will be matched for SFA and dietary cholesterol, but will differ in total fat, primarily MUFA as provided by the avocado. The moderate fat plus avocado diet will provide 34% of calories from total fat, 18% calories from MUFA, and 9% calories from PUFA.
  Interventions: Other: Avocado Diet

INTERVENTIONS:
Other: Avocado Diet — The avocado diet will be designed to ensure that all subjects incorporate 1 avocado (~136g) per day into a moderate fat diet. Both the Lower-Fat diet and avocado diet will be matched for SFA and dietary cholesterol, but will differ in total fat, primarily MUFA as provided by the avocado. The moderate fat plus avocado diet will provide 34% of calories from total fat, 18% calories from MUFA, and 9% calories from PUFA.
  Other Names: moderate fat plus avocado
  Arms: Avocado Diet
Other: Lower-Fat Diet — The Lower-Fat diet will provide ~24% of calories from fat and meet the SFA and cholesterol recommendations of a Step-II diet recommended by the National Heart, Lung, and Blood Association's National Cholesterol Education Program. SFA will provide 7% of calories, and cholesterol will be less than 200mg/day. Vegetables and fruits in the Lower-Fat diet will be selected from foods that are low in antioxidants.
  Other Names: lower-fat,low SFA diet
  Arms: Lower-Fat Diet
Other: Moderate Fat Diet — This diet is designed to be the control diet for the avocado diet and will have an identical fatty acid profile. MUFA-enriched food (fats) will be substituted for avocado. The substitution foods will not contain antioxidant or cholesterol-lowering components similar to those in avocado.
  Other Names: moderate fat without avocado
  Arms: Moderate Fat Diet

SUMMARY:
The investigators propose to evaluate the effects of avocado consumption (by incorporating 1 unit of fruit per day into a healthy diet) on multiple cardiovascular disease (CVD) risk factors. The investigators will compare chronic consumption of a moderate fat blood cholesterol-lowering diet incorporating one avocado per day versus a blood cholesterol-lowering Lower-Fat diet on established CVD risk factors including lipids and lipoproteins, and blood pressure (BP). The investigators also will evaluate the effects of an avocado diet on several emerging CVD risk factors. To elucidate the specific benefits of avocado and its accompanying bioactives on the aforementioned risk factors, the investigators will compare the avocado diet with a diet that has the same macronutrient profile (but without the avocado).

DETAILED DESCRIPTION:
A randomized, 3-period cross-over, controlled feeding study was designed to compare the effects of a moderate fat blood cholesterol-lowering diet that provides one avocado per day (total fat = 34% total energy, MUFA=18%, SFA <7%) to an Average American diet (AAD), Lower-Fat diet (total fat = 24% total energy, SFA <7%), and Moderate Fat diet (with equivalent fatty acid profile to the avocado diet) without avocado. The study population consists of 40 overweight (BMI25-35 kg/m2) men and women with moderately elevated LDL-C, between the25-90th percentiles from NHANES. The investigators hypothesize that a moderate fat heart-healthy diet, including 1 avocado per day will reduce CVD risk factors including lipids, lipoproteins, apolipoproteins, lipoprotein particle size, markers of oxidative stress and inflammation, blood pressure and reverse cholesterol transport compared to an AAD, Lower-Fat diet, and moderate fat diet without avocado.

ELIGIBILITY:
Inclusion Criteria:

* healthy non-smoking
* overweight (BMI 25-35 kg/m2) men and women
* LDL-C between the25-90th percentile from NHANES: 105-194mg/dL for males; 98-190mg/dL for females)

Exclusion Criteria:

* BP >140/90 mmHg;
* A history of myocardial infarction, stroke, diabetes mellitus, liver disease, kidney disease, and thyroid disease (unless controlled on medication);
* Lactation, pregnancy, or desire to become pregnant during the study;
* Cholesterol-lowering medication use;
* Intake of putative cholesterol-lowering supplements (psyllium, fish oil capsules, soy lecithin, niacin, fiber, flax, and phytoestrogens, stanol/sterol supplemented foods);
* Vegetarianism;
* Nut allergies (Other food allergies were reviewed on a case-by-case basis);
* Refusal to discontinue nutritional supplements, herbs or vitamins

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Lipids and lipoproteins | The end of each diet period
  Total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides are measured as part of the lipids and lipoprotein profile.
  Diet period one runs for 5 weeks after a 2-week run-in diet, then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks
Lipoprotein particle size | The end of each diet period
  Advanced lipoprotein testing is used to measure LDL particle size and subclasses of HDL and VLDL.
  Diet period one runs for 5 weeks after a 2-week run-in diet (baseline), then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks

SECONDARY OUTCOMES:
Oxidized-LDL | The end of each diet period
  Diet period one runs for 5 weeks after a 2-week run-in diet, then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks
lipid hydroperoxide | The end of each diet period
  Diet period one runs for 5 weeks after a 2-week run-in diet, then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks
Macrophage Cholesterol efflux | The end of each diet period
  Diet period one runs for 5 weeks after a 2-week run-in diet, then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks
HDL anti-inflammatory function | The end of each diet period
  Diet period one runs for 5 weeks after a 2-week run-in diet, then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks
Serum fatty acid profile | The end of each diet period
  Diet period one runs for 5 weeks after a 2-week run-in diet, then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks
Inflammatory biomarkers | The end of diet period
  CRP and IL-6 are measured as the markers of inflammation.
  Diet period one runs for 5 weeks after a 2-week run-in diet, then there is a 2-3 week compliance break, and then diet period two runs for another 5 weeks; then there is a 2-3 week compliance break, and then diet period three runs for another 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, Dr., Principal Investigator — Penn State University; Li Wang, Study Director — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Tindall AM, Kris-Etherton PM, Petersen KS. Replacing Saturated Fats with Unsaturated Fats from Walnuts or Vegetable Oils Lowers Atherogenic Lipoprotein Classes Without Increasing Lipoprotein(a). J Nutr. 2020 Apr 1;150(4):818-825. doi: 10.1093/jn/nxz313. PMID 31909809
- [Derived] Wang L, Tao L, Hao L, Stanley TH, Huang KH, Lambert JD, Kris-Etherton PM. A Moderate-Fat Diet with One Avocado per Day Increases Plasma Antioxidants and Decreases the Oxidation of Small, Dense LDL in Adults with Overweight and Obesity: A Randomized Controlled Trial. J Nutr. 2020 Feb 1;150(2):276-284. doi: 10.1093/jn/nxz231. PMID 31616932
- [Derived] Wang L, Bordi PL, Fleming JA, Hill AM, Kris-Etherton PM. Effect of a moderate fat diet with and without avocados on lipoprotein particle number, size and subclasses in overweight and obese adults: a randomized, controlled trial. J Am Heart Assoc. 2015 Jan 7;4(1):e001355. doi: 10.1161/JAHA.114.001355. PMID 25567051